CLINICAL TRIAL: NCT06849960
Title: Reliabilitiy and Validity of the Two-minute Step Test in Patients With Multiple Sclerosis
Brief Title: Relıabılıty and valıdıty of the Two-minute Test wıth Multiple Sclerosis
Status: Enrolling by invitation | Type: Observational
Sponsor: Sanko University (Other)
Responsible Party: Principal Investigator, Hakan Polat, Physiotherapy and Rehabilitation Department, Assistant Professor, Sanko University
Other Study IDs: hakanpolatt
Record Dates: First submitted 2025-02-23; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study will include 50 MS patients who were examined by a specialist neurologist diagnosed according to McDonalds criteria in the Neurology Outpatient Clinic of SANKO University Sani Konukoğlu Application and Research Hospital and whose informed consent was obtained. Ethical approval of the study was obtained from SANKO University Non-Interventional Clinical Research Ethics Committee (No:2025/01- ethics committee decision No:2).

MS patients between the ages of 18-65 years, with an Expanded Disability Status Scale (EDSS) score ≤ 4, who are not pregnant, who have not had an attack in the last 1 month and who have not received corticosteroid treatment will be included in the study. Individuals who have taken any medication that may affect walking and balance ability in the last month, have orthopedic, other neurologic diseases and cognitive problems will not be included in the study.

Demographic information (age, height, weight, body mass index and gender) of individuals with MS will be recorded. Firstly, the tests will be explained to the individuals in detail.Assessments will be performed by a physiotherapist with 10 years of experience in this field.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) is a demyelinating, inflammatory, neurodegenerative and progressive disease with a complex etiology. the symptoms of the disease vary according to the lesion site and generally include problems such as balance and fall problems, fatigue, loss of strength and spasticity in the lower extremities, and sensory disturbances.

The study will include 50 MS patients who were examined by a specialist neurologist diagnosed according to McDonalds criteria in the Neurology Outpatient Clinic of SANKO University Sani Konukoğlu Application and Research Hospital and whose informed consent was obtained. Ethical approval of the study was obtained from SANKO University Non-Interventional Clinical Research Ethics Committee (No:2025/01- ethics committee decision No:2).

MS patients between the ages of 18-65 years, with an Expanded Disability Status Scale (EDSS) score ≤ 4, who are not pregnant, who have not had an attack in the last 1 month and who have not received corticosteroid treatment will be included in the study. Individuals who have taken any medication that may affect walking and balance ability in the last month, have orthopedic, other neurologic diseases and cognitive problems will not be included in the study.

Demographic information (age, height, weight, body mass index and gender) of individuals with MS will be recorded. Firstly, the tests will be explained to the individuals in detail.Assessments will be performed by a physiotherapist with 10 years of experience in this field.

Assessments will be performed separately by two physiotherapists on two consecutive days. Each physiotherapist will administer the tests in two separate sessions on one day. The time to complete the activities during the tests will be recorded with a stopwatch. Patients will be unaware of the recorded time. Individuals will be rested before the tests. On the first day, the first assessor will administer the 2MST in the first session. Then 2MWT and Single Leg Stance tests will be performed respectively. In the next session, the second evaluator will perform the 2MST. On the 2nd day of the assessment, the second assessor will first perform the 2MST. Then, the first assessor will perform the 2MST. In both sessions, individuals will be assessed in the same environment to minimize the influence of environmental factors. This environment has adequate lighting and the floor of the room has a hard surface as a safety precaution due to the risk of falling. Due to the risk of heat intolerance problem in MS, attention was paid to the room temperature and the room temperature will be at normal room temperature.

ELIGIBILITY:
Inclusion Criteria:

* being diagnosed with revised 2017 McDonald criteria,
* aged older than 18 years,
* ability to walk with or without aid,
* no medication changes in the last 2 months,
* volunteering to participate in the research,
* not having any obstacles to verbal and cognitive communication.

Exclusion Criteria:

* having orthopedic, psychological, and other neurological disorders, having had -a relapse in the past 3 months
* having pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PATIENTS DIAGNOSED WITH MULTIPLE SCLEROSIS ADMITTED TO THE NEUROLOGY OUTPATIENT CLINIC OF SANKO UNİVERSİTESİ SANİ KONUKOĞLU APPLICATION AND RESEARCH HOSPITA
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-02-15 (Actual); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
2 min step test (2MST) | 1 years
  The 2MST is a test used to measure physical performance. Before starting the test, the wall was marked with tape at the midpoint between the spina iliaca anteriosuperior and the patella. The participant was asked to start walking in place without running when the signal was given. During the test, the number of right and left knee lifts reaching the mark within 2 minutes was recorded . The most affected side's results of patients were used for analysis.
2-min walk test (2MWT) | 1 years
  This test measures the distance that individuals walk in 2 minutes and assesses their functional capacity. The person walks for 2 minutes at maximum speed between two cones placed by measuring 15 meters. If an assistive device is used, the person can walk with the device. Since 6-minute walk test may cause fatigue in MS patients, 2MWT is recommended. Its validity in MS was demonstrated by Scalzitti et al.
One-leg stand test (OLSTS) | 1 years
  OLSTS measured the time that the person could maintain the posture without losing balance in a standing position on one leg with eyes open. It was repeated for both feet. The most affected side's results of patients were used for analysis.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Sanko University, Şehitkamil, Gaziantep
  - Sanko University, Gaziantep, Şehi̇tkami̇l

IPD SHARING:
Plan to Share IPD: Undecided
will be decided when the study is completed

REFERENCES:
- [Result] de Jesus SFC, Bassi-Dibai D, Pontes-Silva A, da Silva de Araujo A, de Freitas Faria Silva S, Veneroso CE, de Paula Gomes CAF, Dibai-Filho AV. Construct validity and reliability of the 2-Minute Step Test (2MST) in individuals with low back pain. BMC Musculoskelet Disord. 2022 Dec 5;23(1):1062. doi: 10.1186/s12891-022-06050-w. PMID 36471309
- [Result] Braghieri HA, Kanegusuku H, Corso SD, Cucato GG, Monteiro F, Wolosker N, Correia MA, Ritti-Dias RM. Validity and reliability of 2-min step test in patients with symptomatic peripheral artery disease. J Vasc Nurs. 2021 Jun;39(2):33-38. doi: 10.1016/j.jvn.2021.02.004. Epub 2021 Mar 19. PMID 34120695
- [Derived] Polat H, Katirci-Kirmaci ZI, Uzun M, Ekmekyapar-Firat Y, Erel S, Neyal AM. Validity, intra-rater and inter-rater reliability, and minimal detectable change of the two-minute step test in patients with multiple sclerosis. Mult Scler Relat Disord. 2025 Dec;104:106773. doi: 10.1016/j.msard.2025.106773. Epub 2025 Sep 19. PMID 41038137